CLINICAL TRIAL: NCT01182350
Title: Phase II Trial of Molecularly Determined Treatment of Children and Young Adults With Newly Diagnosed Diffuse Intrinsic Pontine Gliomas
Brief Title: Molecularly Determined Treatment of Diffuse Intrinsic Pontine Gliomas (DIPG)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per design: Stop if fewer than 3 cohorts by molecular classification were with 10 participants or only 1 cohort enrolled at least 15 participants of 50.
Sponsor: Karen D. Wright MD (Other)
Collaborators: Boston Children's Hospital (Other); University of California, San Francisco (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Healthcare of Atlanta (Other); Children's Hospital Colorado (Other); Children's Hospital Los Angeles (Other); Children's Hospital of Michigan (Other); Children's Hospitals and Clinics of Minnesota (Other); Cook Children's Medical Center (Other); OHSU Doernbecher Children's Hospital (Other); Duke University (Other); Johns Hopkins University (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Nemours Children's Clinic (Other); New York University (Other); Milton S. Hershey Medical Center (Other); Seattle Children's Hospital (Other); Lucile Packard Children's Hospital (Other); University of Louisville (Other); Children's National Research Institute (Other); Washington University School of Medicine (Other); Phoenix Children's Hospital (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor-Investigator, Karen D. Wright MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFCI 10-321
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: Molecularly Determined Treatment
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Bevacizumab; Erlotinib Hydrochloride; Temozolomide; Radiation

STUDY DESIGN:
Intervention Model Description: This is not a randomized trial rather participants are classified and therapy is directed based on molecular profile obtained from surgical biopsy.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- radiation + bevacizumab (Experimental): Cohort 1: MGMT-/EGFR-
  Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Interventions: Drug: Bevacizumab; Radiation: Radiation
- radiation + bevacizumab + erlotinib (Experimental): Cohort 2: MGMT-/EGFR+
  Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Erlotinib: Administered orally at 85 mg/m2 daily continuously during radiation therapy, through the interim period and for up to 10 maintenance cycles
  Interventions: Drug: Bevacizumab; Drug: Erlotinib
- radiation + bevacizumab + temozolomide (Experimental): Cohort 3. MGMT+/EGFR-
  Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Temozolomide: Administered orally at 90 mg/m2/day continuously during radiation therapy, held through the interim period and then 200 mg/m2/day for 5 days for up to 10 maintenance cycles
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Radiation: Radiation
- radiation + bevacizumab + erlotinib + temozolomide (Experimental): Cohort 4. MGMT+/EGFR+
  Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Erlotinib: Administered orally at 85 mg/m2 daily continuously during radiation therapy, through the interim period and for up to 10 maintenance cycles
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Temozolomide; Radiation: Radiation

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
Drug: Erlotinib
  Other Names: Tarceva
  Arms: radiation + bevacizumab + erlotinib; radiation + bevacizumab + erlotinib + temozolomide
Drug: Temozolomide
  Other Names: Temodar
  Arms: radiation + bevacizumab + erlotinib + temozolomide; radiation + bevacizumab + temozolomide
Radiation: Radiation
  Other Names: irradiation
  Arms: radiation + bevacizumab; radiation + bevacizumab + erlotinib + temozolomide; radiation + bevacizumab + temozolomide

SUMMARY:
Diagnosis of diffuse intrinsic pontine glioma (DIPG) for decades has relied on imaging studies and clinical findings. Histologic confirmation has been absent with surgical biopsy of brainstem tumors not believed to have acceptable safety. The prognosis of DIPG has remained quite poor and novel therapeutic strategies are needed. This DIPG Biology and Treatment Study (DIPG-BATS) study incorporates a surgical biopsy at presentation using strict preoperative neurosurgical planning and stratifies participants to receive FDA-approved agents chosen on the basis of specific biologic targets. This is the first prospective national clinical trial to examine the feasibility and safety of incorporating surgical biopsy into potential treatment strategies for children with DIPG.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the overall survival of children and young adults with DIPG in the context of a molecularly based treatment strategy, compared to historical controls (COG ACNS0126). Secondary objectives were to determine the safety and potential morbidity associated with biopsy of classic DIPGs based on imaging and clinical history as well as ability to perform biologic analyses on the biopsy material obtained to guide therapy. At study entry, a MRI-guided frameless or frame-based stereotactic biopsy will be performed approaching the pontine termentum through a trans-cerebellar or trans-frontal route. The exact biopsy location will be determined by the treating neurosurgeon at the designated participating site with the goal of minimizing procedural risk. Treatment directed based on tumor biopsy results requires classification of patients into 1 of 4 potential cohorts: O^6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status (negative versus positive) and epidermal growth factor receptor (EGFR) overexpression status (negative versus positive).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

1. Tumor: Newly diagnosed non-disseminated diffuse intrinsic pontine glioma based on classic clinical AND radiographic finding.
2. No prior radiation therapy or chemotherapy.
3. Age: Patient must be 3 to < 18 years of age at the time of diagnosis.
4. Performance Score: Karnofsky Performance Scale > 12 y/o >/= 50 or Lansky Performance Score for patients < 12y/o 50 assessed within two-weeks prior to enrollment.
5. Participants must have normal organ and marrow function as defined below within two week s prior to enrollment:

   * Absolute neutrophil count > 1,000/mcL
   * Platelets > 100,000/mcL (transfusion independent)
   * Hemoglobin > 8gm/dL (can be transfused)
   * Hepatic: Total bilirubin < 1.5 times the upper limit of normal; alanine aminotransferase [SGPT (ALT)] and aspartate aminotransferase [SGOT (AST)] < 5 times the institutional upper limit of normal.
   * Renal: Serum creatinine which is less than 1.5x the upper limit of institutional normal for age or Glomerular Filtration Rate (GFR) > 70 ml/min/1.73m2.
6. Female patients of childbearing potential must have negative serum or urine pregnancy test. Patient must not be pregnant or breast feeding.
7. Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
2. Patients receiving any other anticancer or experimental drug therapy.
3. Patients with disseminated intrinsic diffuse brainstem gliomas in either brain or spine (can be based on clinical evaluation).
4. Participants receiving any medications or substances that are strong/intermediate inhibitors or inducers of Cytochrome P450 (CYP450), Cytochrome P3A4(CYP3A4) or Cytochrome 1A2 (CYP1A2) are ineligible. Lists including medications and substances known or with the potential to interact with the CYP450 CYP3A4 or CYP1A2 isoenzymes are provided in Appendix I.
5. Use of hematopoietic growth factors within the 2 weeks prior to initiation of therapy.
6. Patients with evidence of spontaneous hemorrhage greater than 0.5cm unrelated to surgery.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Pregnant women are excluded from this study because bevacizumab, temozolomide and erlotinib can have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued.

   -

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen D. Wright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (23):
- United States (23):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University/Lucile Packard Children's Hospital, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta N, Goumnerova LC, Manley P, Chi SN, Neuberg D, Puligandla M, Fangusaro J, Goldman S, Tomita T, Alden T, DiPatri A, Rubin JB, Gauvain K, Limbrick D, Leonard J, Geyer JR, Leary S, Browd S, Wang Z, Sood S, Bendel A, Nagib M, Gardner S, Karajannis MA, Harter D, Ayyanar K, Gump W, Bowers DC, Weprin B, MacDonald TJ, Aguilera D, Brahma B, Robison NJ, Kiehna E, Krieger M, Sandler E, Aldana P, Khatib Z, Ragheb J, Bhatia S, Mueller S, Banerjee A, Bredlau AL, Gururangan S, Fuchs H, Cohen KJ, Jallo G, Dorris K, Handler M, Comito M, Dias M, Nazemi K, Baird L, Murray J, Lindeman N, Hornick JL, Malkin H, Sinai C, Greenspan L, Wright KD, Prados M, Bandopadhayay P, Ligon KL, Kieran MW. Prospective feasibility and safety assessment of surgical biopsy for patients with newly diagnosed diffuse intrinsic pontine glioma. Neuro Oncol. 2018 Oct 9;20(11):1547-1555. doi: 10.1093/neuonc/noy070. PMID 29741745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study screening procedures were conducted at 23 sites in the United States. Eligible participants enrolled between September 2011 and September 2015.
Groups:
- Cohort 1: MGMT-/EGFR-; Cohort 2: MGMT-/EGFR+: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
- Cohort 3 MGMT+/EGFR-: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles Temozolomide: Administered orally at 90 mg/m2/day continuously during radiation therapy, held through the interim period and then 200 mg/m2/day for 5 days for up to 10 maintenance cycles
- Cohort 4. MGMT+/EGFR+: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles Erlotinib: Administered orally at 85 mg/m2 daily continuously during radiation therapy, through the interim period and for up to 10 maintenance cycles
  Temozolomide: Administered orally at 90 mg/m2/day continuously during radiation therapy, held through the interim period and then 200 mg/m2/day for 5 days for up to 10 maintenance cycles
- Ineligible for Direct Treatment Assignment: All enrolled participants were to receive surgical biopsy to guide treatment assignment based on molecular results.Participants without an evaluable sample were ineligible for direct treatment assignment.
Period: Overall Study
Arm/Group | Cohort 1: MGMT-/EGFR- | Cohort 2: MGMT-/EGFR+ | Cohort 3 MGMT+/EGFR- | Cohort 4. MGMT+/EGFR+ | Ineligible for Direct Treatment Assignment
Started | 30 | 14 | 3 | 3 | 3
Underwent Stereotactic Biopsy | 30 | 14 | 3 | 3 | 0
Started Assigned Chemoradiation | 27 | 14 | 2 | 2 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 27 | 14 | 3 | 3 | 3
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 15 | 12 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 1 | 0
Not completed — Alternative Therapy | 2 | 0 | 1 | 0 | 0
Not completed — Travel Issue/Prefer Treatment at Home | 2 | 0 | 1 | 1 | 0
Not completed — Unevaluable for Biopsy | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants who underwent stereotactic biopsy.
Groups:
- All Biopsied Participants: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Treatment directed based on tumor biopsy results requires classification of patients into 1 of 4 potential cohorts: O^6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status (negative versus positive) and epidermal growth factor receptor (EGFR) overexpression status (negative versus positive).
Arm/Group | All Biopsied Participants
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 6.3 [3.3 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Molecular Classification [Count of Participants; unit: Participants] — Treatment directed based on tumor biopsy results requires classification of patients into 1 of 4 potential cohorts: O^6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status (negative versus positive) and epidermal growth factor receptor (EGFR) overexpression status (negative versus positive).
  Participants
    MGMT-/EGFR- | 30
    MGMT-/EGFR+ | 14
    MGMT+/EGFR- | 3
    MGMT+/EGFR+ | 3

OUTCOME MEASURES:

1. Primary Outcome: 9-month Overall Survival (OS) Rate
Description: 9-month overall survival is the percentage of participants remaining alive 9 months from registration.
Time Frame: 9 months
Population: The analysis population is comprised of the subset of participants who underwent biopsy, obtained a molecularly-based treatment assignment and started assigned chemoradiation therapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Patients Starting Assigned Chemoradiation: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Treatment directed based on tumor biopsy results requires classification of patients into 1 of 4 potential cohorts: O^6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status (negative versus positive) and epidermal growth factor receptor (EGFR) overexpression status (negative versus positive).
Arm/Group | All Patients Starting Assigned Chemoradiation
Number analyzed (Participants) | 45
percentage of participants | 64.4 [51.1 to 76.3]

2. Secondary Outcome: Rate of Lethal Complications From Surgery
Description: The rate of lethal complications from surgery is the percentage of participants dying as a result of surgery.
Time Frame: 2 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Biopsied Participants: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Treatment directed based on tumor biopsy results requires classification of patients into 1 of 4 potential cohorts: O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status (negative versus positive) and epidermal growth factor receptor (EGFR) overexpression status (negative versus positive).
Arm/Group | All Biopsied Participants
Number analyzed (Participants) | 50
percentage of participants | 0.0 [0.0 to 5.8]

3. Secondary Outcome: Grade 3-4 Post-Procedural Surgery-Related Toxicity Rate
Description: Grade 3-4 post-procedural surgery-related toxicity rate is the percentage of participants experiencing at least one grade 3-4 adverse event (AE) during the post-procedural time frame of 14 days attributable to the surgical procedure based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4).
Time Frame: 2 weeks
Population: The analysis dataset is comprised of all enrolled participants who underwent stereotactic biopsy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Biopsied Participants
Number analyzed (Participants) | 50
percentage of participants | 10.0 [4.1 to 19.9]

4. Secondary Outcome: Delay in Radiation Therapy Start
Description: The number of participants delaying the start of radiation therapy by more than 3 weeks due to complications as a result of surgical biopsy to obtain diagnostic tumor sample.
Time Frame: 3 weeks
Population: The analysis dataset is comprised of all enrolled participants who underwent stereotactic biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | All Biopsied Participants
Number analyzed (Participants) | 50
Participants | 1

5. Secondary Outcome: Feasibility Rate of Molecular Approach to Therapy
Description: Feasibility rate of the molecular strategy is based on the percentage of participants either with inadequate tissue from surgical biopsy to confirm DIPG diagnosis and/or with uninterpretable results for identification of EGFR overexpression and MGMT methylation status.
Time Frame: 3 weeks
Population: The analysis dataset is comprised of all enrolled participants who underwent stereotactic biopsy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Biopsied Participants
Number analyzed (Participants) | 50
percentage of participants | 92.0 [82.6 to 97.2]

6. Secondary Outcome: Number of Participants With Grade 3-4 Treatment-Related Toxicity Over Chemoradiation Therapy
Description: Counts any participant experiencing at least one treatment-related grade 3 or 4 adverse event (AE) with treatment attribution of possibly, probably or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) over chemoradiation therapy as reported on case report forms.
Time Frame: Adverse events were routinely throughout treatment. Treatment duration was a median of 6.4 months (range 0.4-13.4 months) in this study cohort.
Population: The analysis population is comprised of the subset of participants who underwent surgical biopsy, obtained a molecularly-based treatment assignment and started assigned chemoradiation therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 MGMT-/EGFR-: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
- Cohort 2 MGMT-/EGFR+: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles Erlotinib: Administered orally at 85 mg/m2 daily continuously during radiation therapy, through the interim period and for up to 10 maintenance cycles
- Cohort 3: MGMT+/EGFR-: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles Temozolomide: Administered orally at 90 mg/m2/day continuously during radiation therapy, held through the interim period and then 200 mg/m2/day for 5 days for up to 10 maintenance cycles
Arm/Group | Cohort 1 MGMT-/EGFR- | Cohort 2 MGMT-/EGFR+ | Cohort 3: MGMT+/EGFR- | Cohort 4. MGMT+/EGFR+
Number analyzed (Participants) | 27 | 14 | 2 | 2
Participants | 5 | 5 | 0 | 0

7. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration of time [months (m)] from study entry to documented disease progression (PD) or death. Participants alive without PD are censored at the date of last disease assessment. For intrinsic pontine brainstem gliomas, only one lesion/mass is present at diagnosis. Comparisons of maximal 2-dimensional measurements, TxW (product of the longest diameter [width (W)] and its longest perpendicular diameter [transverse (T)]) are used to assess response for this target lesion. PD is 25% or more increase, taking as reference the smallest product observed since the start of treatment, or the appearance of one or more new lesions.
Time Frame: Disease assessments using a standard CNS imaging protocol occurred chemoradiation cycles 1 and 2, every other maintenance cycle, every 3 months post-treatment year 1 then annually until PD or therapy change; In this study cohort, follow-up was up to 34m.
Population: The analysis population is comprised of the subset of participants who underwent surgical biopsy, obtained a molecularly-based treatment assignment and started assigned chemoradiation therapy. The PFS was aggregated across cohorts per statistical analysis plan to evaluate the effect of the "molecular strategy".
Measure: Median (Full Range); unit: months
Arm/Group | All Patients Starting Assigned Chemoradiation
Number analyzed (Participants) | 45
months | 8 [1 to 16]

8. Post Hoc Outcome: 9-month Overall Survival (OS) Rate by Molecular Cohort
Description: 9-month OS rate is the percentage of participants alive at 9 months from registration.
Time Frame: 9 months
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2: MGMT-/EGFR+; Cohort 4. MGMT+/EGFR+: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Erlotinib: Administered orally at 85 mg/m2 daily continuously during radiation therapy, through the interim period and for up to 10 maintenance cycles
- Cohort 3. MGMT+/EGFR-: Protocol treatment lasts approximately 52 weeks including a 4-week interim period once radiation therapy is completed and a maintenance phase (cycle duration=28 days).
  Radiation therapy: Given in 180 cGy fractions to a total dose of 59.4 + 1.8 Gy/-5.4 Gy for approximately 7 weeks beginning 7-21 days after biopsy
  Bevacizumab: Administered intravenously at 10 mg/kg beginning no sooner than 21 days from biopsy and every 14 days concurrent with radiation therapy, through the interim period and for up to 10 maintenance cycles
  Temozolomide: Administered orally at 90 mg/m2/day continuously during radiation therapy, held through the interim period and then 200 mg/m2/day for 5 days for up to 10 maintenance cycles
Arm/Group | Cohort 1: MGMT-/EGFR- | Cohort 2: MGMT-/EGFR+ | Cohort 3. MGMT+/EGFR- | Cohort 4. MGMT+/EGFR+
Number analyzed (Participants) | 27 | 14 | 2 | 2
percentage of participants | 66.7 [49.1 to 81.4] | 57.1 [32.5 to 79.4] | 50.0 [2.6 to 97.5] | 100 [22.4 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were routinely throughout treatment. Treatment duration was a median of 6.4 months (range 0.4-13.4 months) in this study cohort.
Description: Maximum grade toxicity by type was first calculated within each arm. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term. The analysis population is comprised of the subset of participants who underwent surgical biopsy.
Arm/Group | Cohort 1 MGMT-/EGFR- | Cohort 2 MGMT-/EGFR+ | Cohort 3: MGMT+/EGFR- | Cohort 4. MGMT+/EGFR+
All-Cause Mortality (participants affected / at risk) | 29/30 | 14/14 | 3/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 8/30 | 9/14 | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 30/30 | 14/14 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 MGMT-/EGFR- (N=30) | Cohort 2 MGMT-/EGFR+ (N=14) | Cohort 3: MGMT+/EGFR- (N=3) | Cohort 4. MGMT+/EGFR+ (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dysphasia (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 2 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Spasticity (Nervous system disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 MGMT-/EGFR- (N=30) | Cohort 2 MGMT-/EGFR+ (N=14) | Cohort 3: MGMT+/EGFR- (N=3) | Cohort 4. MGMT+/EGFR+ (N=3)
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 1 | 0
Abducens nerve disorder (Nervous system disorders) | 6 | 4 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 10 | 6 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 4 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 5 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 5 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 7 | 4 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cardiac disorders - Other (Cardiac disorders) | 1 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 11 | 5 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 2 | 1
Creatinine increased (Investigations) | 1 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 5 | 3 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Death NOS (General disorders) | 2 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 3 | 1 | 1 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 6 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 8 | 0 | 1
Dysarthria (Nervous system disorders) | 3 | 3 | 1 | 0
Dysesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Dysphasia (Nervous system disorders) | 2 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 0
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 0 | 0
Encephalitis infection (Infections and infestations) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eye disorders - Other (Eye disorders) | 7 | 2 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 1 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 6 | 3 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1
Fatigue (General disorders) | 14 | 4 | 1 | 1
Fever (General disorders) | 4 | 4 | 1 | 1
Flushing (Vascular disorders) | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 4 | 3 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Glossopharyngeal nerve disorder (Nervous system disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 20 | 7 | 2 | 0
Hemoglobin increased (Investigations) | 2 | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 3 | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 5 | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 16 | 6 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 5 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 0
Hypoglossal nerve disorder (Nervous system disorders) | 2 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3 | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 4 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 3 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 3 | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 5 | 0 | 2 | 1
Investigations - Other (Investigations) | 0 | 2 | 0 | 1
Irritability (General disorders) | 4 | 2 | 0 | 0
IVth nerve disorder (Nervous system disorders) | 2 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 16 | 5 | 1 | 1
Malaise (General disorders) | 1 | 2 | 0 | 0
Mediastinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 5 | 3 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 4 | 2 | 3
Neck edema (General disorders) | 0 | 1 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 4 | 3 | 1 | 1
Neutrophil count decreased (Investigations) | 5 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 3 | 1 | 0 | 0
Oculomotor nerve disorder (Nervous system disorders) | 3 | 1 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pain (General disorders) | 5 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 2 | 0 | 0
Platelet count decreased (Investigations) | 10 | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 4 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 2 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 2
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 1 | 0 | 0
Salivary gland fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 6 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Spasticity (Nervous system disorders) | 2 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 2 | 0 | 0
Upper respiratory infection (Infections and infestations) | 7 | 4 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 5 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Vagus nerve disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 16 | 9 | 1 | 3
Weight gain (Investigations) | 6 | 4 | 1 | 0
Weight loss (Investigations) | 3 | 3 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
White blood cell decreased (Investigations) | 13 | 3 | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early having met the pre-specified stopping rule which required 3 or more cohorts with at least 10 patients each or 2 cohorts with at least 15 patients each in the first 50 patients with informative biopsies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No